CLINICAL TRIAL: NCT04338789
Title: Mandibular Molar Protraction Assisted by Temporary Anchorage Device and Piezoelectric Corticotomy
Brief Title: Accelerated Mandibular Molar Protraction: Piezocision at the Time of Molar Protraction or Later?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Elham Abu Alhaija, Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 266/216
Record Dates: First submitted 2020-02-25; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Orthodontic Appliance
Keywords: Piezocision; molar protraction; Accelerated

STUDY DESIGN:
Intervention Model Description: Split mouth design where piezocision will be performed at the time of molar protraction on the right or left side of the bilateral first molar extraction subjects and 3 months of molar protraction on the other side. A third group of subjects will act as a control where molar protraction will be done with no piezocision.
  - Comparison between the 3 groups of subjects; Early piezocision, late piezocision and no piezocision molar protraction groups.
Who Masked: Outcomes Assessor
Masking Description: Blinding of either patient or clinician was not possible during treatment. However, partial blinding was possible. Orthodontic molar protraction was carried out by the clinician without knowing the GCF levels and the lab was blinded to the clinical findings. Also, periapical radiographs and study casts were masks during data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): It consisted of 20 subjects with bilateral first molar extraction space where piezocesion was performed immediately before molar protraction on the left or right side of the patient.
  Interventions: Other: Piezocision
- Group 2 (Experimental): It consisted of 20 subjects with bilateral first molar extraction space where piezocesion was performed 3 months after molar protraction with no piezocision on the left or right side of the patient.
  Interventions: Other: Piezocision
- Group 3 (No Intervention): It consisted of 20 subjects (40 molars) where molar protraction was performed with no piezocesion.

INTERVENTIONS:
Other: Piezocision — Piezocesion was performed by making 2 vertical incisions mesial and distal to the extraction space. Piezotome was inserted in the incisions previously made and bone cuts were done with a length up to mucogingival line and depth of 3 mm.
  Arms: Group 1; Group 2

SUMMARY:
This study was conducted to compare the rate of second molar protraction, level of Interleukin1-β in gingival crevicular fluid, periodontal health (gingival index, plaque index, and periodontal pocket depth) and root resorption in patients treated by molar protraction with piezocision performed early at the time of protraction (Group 1), piezocision performed 3 months after molar protraction (Group 2), and no piezocision molar protraction (Group 3).

DETAILED DESCRIPTION:
Detailed Description: Thirty-five subjects who presented with bilaterally extracted mandibular first molar were selected to participate in the study. The subjects were subdivided into one of 3 groups as follows: group 1 consisted of 20 subjects /20 molars where piezocision was performed immediately before molar protraction; group 2 consisted of 20 subjects/ 20 molars where molar protraction was carried on after 3 months of molar protraction with no piezocision; group 3 consisted of 20 subjects (40 molars) where protraction was carried out with no piezocision.

After reaching 0.019X0.025" SS arch wire, NiTi coil spring was used for space closure (protraction force was 150g) attached from the lower second molar hook to the head of the mini-screw. Piezocision was performed by making 2 vertical incisions mesial and distal to the extraction space. Piezotome was inserted in the incisions previously made and bone cuts were done with a length up to mucogingival line and depth of 3 mm. Gingival crevicular fluid (GCF) sample was obtained from the mesiogingival side of the lower second permanent molar with use of Periopaper. GCF sample was repeated 1 day, 1 week and 4 weeks after molar protraction with piezocision or with no piezocision. Periodontal parameters were measured and lower molar root resorption was assessed using Perapical radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 19 to 30 years
* Bilaterally extracted mandibular first molar (first molar extracted more than one year ago and with a residual extraction space of more than 6 mm).
* Class 1 malocclusion where molar protraction is indicated.
* All permanent teeth are present except for the extracted mandibular first molars.
* Healthy periodontium (gingival index score ≤ 2, plaque index score ≤ 2 and probing depth < 4mm)

Exclusion Criteria:

* Previous orthodontic treatment
* Any systemic disease
* Smoker
* Poor Oral hygiene

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of molar protraction | 1 year
  Measured in mm/month from dental casts
Changes in the level of of Interleukin1-β | 4 weeks
  Detected in Gingival crevicular fluid (GCF). The periopaper was placed for 60 seconds in the mesiogingival sulcus of the lower second permanent molar and was transferred to an Eppendorf tube containing phosphate buffered saline.

SECONDARY OUTCOMES:
Periodontal parameters (Plaque, gingival health, periodontal pocket depth, alveolar bone height) | 1 year
  Plaque and gingival health are measured using plaque index and gingival index. pocket depth and alveolar height are measured in mm.
Lower molar root resorption | 1 year
  Length of lower second molar roots in mm

CONTACTS AND LOCATIONS:
Overall Officials: Elham S A Alhaija, PhD, Principal Investigator — Prof.

IPD SHARING:
Plan to Share IPD: Undecided